CLINICAL TRIAL: NCT04255290
Title: Efficacy of Plyometric and Eccentric Training in Improving the Strength, Stability and Ability of Women Soccer Players. A Randomized Pilot Study.
Brief Title: Plyometric and Eccentric Training in Improving the Strength, Stability and Ability of Women Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAM-EXPL
Record Dates: First submitted 2020-02-01; First posted 2020-02-05 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Female Athlete
Keywords: Isquiotibial; Plyometrics; Eccentric; Soccer; Prevention
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Leg Squat Lounge: The player will be placed in squat position and her partner will be placed behind, suspending the most posterior leg in the air. With the leg that is supported, you will perform a monopodal jump with controlled fall, supporting the foot from tip to heel. It will be done with both lower limbs performing 1 series of 5 repetitions with 30 seconds of rest between sets. 180 jump: The footballer will start in bipodal support, with the trunk erect and hands on the hips. Perform a bipodal jump with a 180º turn during this, keeping the fall for 2 seconds. Each repetition, the turn will be done in a different sense. It will carry out 2 series of 20 sec of execution with 20 sec of rest between series. Brad jump stick landing: The player will stand in hands-free standing. Perform a bipodal jump as far as possible. The knees will not exceed the tip of the foot and the fall will be with a trunk position as straight as possible. He will make 5 jumps the first two weeks.
  Interventions: Other: Leg Squat Lounge
- Control group (Active Comparator): Nordic Funds: One player will stand on her knees, while the other, behind, fixes her legs. The kneeling footballer must drop forward in a controlled manner until she touches the ground and returns to the starting position. The Diver: Player in monopodal support on the lower limb to work, performing hip flexion with the arms forward and the opposite lower limb back, looking for a horizontality in the pelvis (with 10º-20º knee flexion) It will be done with both lower limbs.
  The Glider: With the footballer standing in front of her partner, holding both of them by the shoulders, she lets one leg slide back while the other stays fixed. To return to the starting position, it will be helped by the other player, while the knee will not exceed 10 degrees of flexion. The distribution of all the exercises will be: 2 sets of 5 repetitions with 20 sec rest between sets
  Interventions: Other: Control group

INTERVENTIONS:
Other: Leg Squat Lounge — The players assigned to the experimental group will receive an intervention through plyometric and eccentric hamstring exercises
  Arms: Experimental group
Other: Control group — The subjects included in the control group will perform an eccentric work protocol
  Arms: Control group

SUMMARY:
Introduction. The high rate of recurrence and clinical involvement of muscle injuries in lower limbs, makes the hamstring musculature a very important structure in the development of athletes. Excentric movements, where eccentric force and flexibility are fundamental, and the quadriceps-hamstrings contraction cycle are risk factors for hamstring muscle injury.

Aim. ascertain the effectiveness of plyometric and excéntric exercises in the improvement of hamstring strength.

Study design. Randomized, prospective, multicenter, single-blind clinical study with athletes.

Methods. This study will be carried out with a sample of 40 women, federated players from 18 to 30 years old. They will be randomized into two groups: experimental (plyometric work and eccentric exercises) and control (eccentric exercises). The intervention will last 6 weeks in which, before each training, they will carry out the intervention, for 20 minutes, 3 days a week. An inter-judges piloting will be carried out. We will analyze the normality of the sample with the Kolmogorov-smirnov test and for the inferential analysis, we will use the t-student test of paired data to observe the difference between each evaluation in each study group, and the repeated measures ANOVA to calculate the effect intra and intergroup. Using Cohen's formula we will calculate the size of the effect.

Expected results. The eccentric work along with the plyometrics improves strength in hamstrings, jumping and stability.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18 to 30 years old
* With 3 or less days of training a week
* Federate in the Community of Madrid (Spain)

Exclusion Criteria:

* Players who are injured and cannot do the job at the time of the study
* Soccer players who have had a hamstring injury in the last 6 months
* To practice another sport
* They are receiving physiotherapy treatment in the lower limb
* Not signing the informed consent document

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline hamstring strength after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The mobile application "Nordic" will be used to assess the strength of the hamstring muscles. With the athlete kneeling on the floor, fixed by a partner from the ankles, she will drop down forward. The evaluator will be on the side, recording with a smartphone (Iphone 7) to measure the moment when the subject uncrosses the arms. The test will be carried out up to three times, taking the measures of the angle of rupture in the exercise (angle that forms the trunk with the ground considering the position of the tibiae). The unit of measure the breaking angle.

SECONDARY OUTCOMES:
Change from baseline the jump after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  With the mobile application "My jump 2.0" the jump will be measured. The athlete will be located 1.5 meters from the evaluator, who will be in front of her with a mobile (iPhone 7 model) at ground level. The test will consist of the realization of a Counter Movement Jump (CMJ). The unit of measure of the jump of the application will be the Newton.
Change from baseline lower limb stability after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  With the Y-Balance test the lower limb stability will be measured. The player will be placed in the center of an inverted Y-shaped figure, and in monopodal support on the leg to be evaluated. 3 attempts will be made for each of the scopes (anterior, posteromedial and posterolateral). The distance will be measured in centimeters, taking as value the arithmetic mean of the three attempts made in each range. The Y-shaped figure will be made with tape on the floor. The distance calculation will be carried out with a tape measure.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- European University of Madrid, Madrid, Spain